CLINICAL TRIAL: NCT02710812
Title: Rectal Sparing Approach After Preoperative Radio and/or Chemotherapy in Patients With Rectal Cancer
Acronym: ReSARCh
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Padova (Other)
Collaborators: Istituto Oncologico Veneto IRCCS (Other); Centro di Riferimento Oncologico - Aviano (Other); Istituto Nazionale per lo Studio e la Cura dei Tumori (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Azienda Ospedaliero, Universitaria Ospedali Riuniti (Other)
Responsible Party: Principal Investigator, Pucciarelli Salvatore, Associate Professor, University of Padova
Other Study IDs: 3554/AO/15
Record Dates: First submitted 2016-03-04; First posted 2016-03-17 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Rectal Neoplasms
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rectum sparing group: Patients who have all of the following requirements:
  1. Major or complete clinical response at restaging after 7-8 weeks from the end of neoadjuvant therapy, confirmed at second restaging (after 11-12 weeks from the end of neoadjuvant therapy);
  2. Written informed consent (after 2nd restaging).
  Note: They will be subject to wait-and-see approach only patients with cCR.
  Interventions: Procedure: Local Excision or Wait-and-See

INTERVENTIONS:
Procedure: Local Excision or Wait-and-See — Local excision can be done both with traditional technique and with endoscopic technique (TEM, TAMIS, etc.).
  The following principles should be respected:
  1. A gross margin of at least 0.5 cm;
  2. full-thickness excision including mucosa, submucosa, muscle and peri-rectal fat;
  3. determination of the specimen on the support by pins at the edges in order to facilitate the interpretation of histological pathologist.

SUMMARY:
The proposed study is an observational, prospective, multicenter study of patients undergoing neoadjuvant therapy for medium-low rectal cancer.

Recently the investigators have published the findings of a multicenter Italian phase II study showing that the rate of local recurrence, with a 3 year follow-up, is less than 5% in patients with baseline T2-3 mid-low rectal cancer who, after preoperative chemoradiotherapy (pCRT), showed a major clinical response and underwent a transanal local excision. Based on these results, an organ-sparing approach for patients showing a major clinical response is feasible without reducing the good results obtained with the standard treatment. While a phase III trial is the best way to compare the standard treatment with the organ-sparing approach (local excision or wait-and-see) it is impracticable and likely unethical. An observational study is therefore one of the best way to evaluate the impact that an organ-sparing approach may have on oncological outcomes, quality of life, and bowel function for patients with rectal cancer who, after a pCRT, show a clinical major/complete response.

This phase II trial is designed to test the hypothesis that conservative treatments, in patients with low-mid rectal cancer who undergo a major or complete clinical response after neoadjuvant treatment, will be safe and effective compared to standard surgery.

The investigators will compare rectum-sparing approaches to standard surgery, firstly in terms of rate of organ preservation at 2 years. Additionally they will compare survival outcomes (DFS, OS), stoma rates, clinical and tumor factors related to pathological complete response, correlation between major and complete clinical response.

To add value, the investigators will measure QoL in patients treated with rectum-sparing approaches in comparison to patients treated with standard surgery (TME or abdomino-perineal amputation).

Rectum-sparing approach can be considered clinically acceptable if percentage of conservation of the rectum at two years is not less than 50%.

The collected data on 164 patients who underwent "rectum-sparing" allow to test the hypothesis that the rectum is preserved in 60% of patients with 80% power (exact binomial test for proportions, alpha = 5 %, 1 tail) and the study will be considered positive if it obtains a frequency of conservation of the rectum of not less than 87 cases.

The analysis results will be reported in accordance with STROBE guidelines (von Elm et al., 2008). For all analyzes, continuous variables are described using the mean and standard deviation of position and appropriate measures when appropriate. Categorical variables will be described using the contingency tables.

DETAILED DESCRIPTION:
Introduction and rationale Neoadjuvant therapy, especially preoperative chemoradiotherapy (pCRT) and short-course radiotherapy followed by total mesorectal excision (TME), is the standard of treatment for mid-low rectal cancer. This approach significantly reduces the rate of local recurrence compared with surgery alone, with post-operative radiochemotherapy or with long-course radiotherapy alone.

Concerning the indication to neoadjuvant treatment and its regimen, there is still a wide discrepancy in the literature. Based on the dutch TME trial, showing a low rate of local recurrence in patients treated with short-course radiotherapy (RT) compared to TME alone, the neoadjuvant therapy indication for rectal cancer was RT short-course alone. Meanwhile, with German trial publication, the indication for rectal cancer treatment, up to 15 cm from anal verge, was combination between hyperfractionated RT and 5-fluorouracil based chemotherapy (CT). Two subsequent trials (Polish trial and Trans-Tasman Radiation Oncology Group trial) showed that RT short-course alone and CRT with hyperfractionated RT have similar oncological outcomes. Thus, in recent years there has been an increasing interest in the administration of neoadjuvant chemotherapy at therapeutic doses and not only radiosensitizers. Regimens are basically as follows: induction regimen and consolidation regimen. In the first case, CT precedes pCRT, while in consolidation regimen CT follows pCRT. The rationale for this strategy is that, currently, the mortality of rectal cancer comes from distant metastases and, given that only a full dose chemotherapy can prevent the occurrence of distant recurrence, the rationale for having chemotherapy as early as possible and in as many patients is feasible (patient compliance performing adjuvant chemotherapy is low, often for complications arising from surgery). More recently, studies have been published on the use of neoadjuvant chemotherapy alone and is currently underway in the US the PROSPECT trial evaluating the possibility of using the only neoadjuvant chemotherapy in selected cases instead of the classic CRT. For many reasons (enrolment of patients in clinical trials, refusal of patients to perform treatments considered standard and toxicity from radio and/or chemotherapy) is not uncommon in clinical practice to observe patients who performed unconventional treatments and not provided by any national or international guideline.

Positive and negative consequences of neoadjuvant treatment Neoadjuvant treatment followed by TME involve a high percentage of side effects associated with surgical complications both early and late, the toxicity associated with radiation or chemotherapy and alteration of bowel function, sexual, fecal continence and thus the quality of life (QoL). Among the advantages of neoadjuvant therapy, particularly the treatment associated CRT, it is notable that in 15-20% of cases have the disappearance of the primary tumor, or a pathologic complete response (pCR). Also lengthening the interval between pRT and/or CT and surgery is associated with an increased rate of pCR, therefore, unlike traditional 4-6 week intervals between the end of neoadjuvant therapy and surgery, currently there is tendency to perform surgery after 8-10 weeks, or even after 12 weeks. In patients with a pCR after neoadjuvant therapy, it have been showed a better outcome in long term than those who have a residual disease.

Rationale behind the rectum-sparing approach In order to avoid the morbidity and functional sequelae associated with neoadjuvant therapy followed by TME and based on excellent outcomes seen in patients with a pCR, it has been proposed that, in patients with a major clinical (mCR) or complete (cCR) response, you can opt for a conservative approach that includes preservation of the rectum. During recent years we are seeing a growing interest in these conservative approaches, as demonstrated by the increasing number of publications on this new therapeutic strategy that includes observation ("wait and see" policy) and local excision.

Local excision. LE is considered essentially an excisional biopsy and the decision to observe the patient (only follow-up) or run a TME after LE depends on the histologic features. Patients with no neoplasia (pCR) or with minimal residual disease (ypT1 with tumor regression grade <3 margins and free) are followed with close follow-up. In the remaining cases it opts for a subsequent intervention of TME. Studies concerning LE after neoadjuvant treatment are numerous with the principal lack is to be retrospective, with a low number and definition is not always clear and concordant for mCR and cCR. In addition, all these studies include patients who can not be subjected to radical surgery due to medical comorbidities or who reject the radical surgical treatment, especially when it is expected the final packaging of a stoma. More recently were published prospective studies both phase 2 and phase 3 that have consistently shown that LE is a feasible approach with oncological results comparable to the standard approach.

Among these studies, it is worth highlighting the presence of a multicenter Italian Phase 2 (Pucciarelli et al, 2013). The authors have shown that the rate of local recurrence, with a median follow-up of 3 years, is less than 5% in patients with cancer of the rectum medium-low cT2-3 that, after pRT and/or CT, have reported a major clinical response and were then subjected to LE. The study was approved by the Ethics Committee of Padua and later by the ethics committees of the other three participating centers. The indications to LE of this new trials are the same as in the previous study.

Wait-and-see. This second approach was designed and developed in Brazil, but it is widely spread throughout the world.

Compared to EL, this approach avoids the entire operation and consequently complications related to LE. However, while LE appears indicated in all patients with cCR and mCR, wait-and-see approach is required when there is a cCR. The reason for the different indication is that the probability that there is a correlation between cCR and pCR is very high; unlike the correlation between mCR and pCR it is much lower. As shown by scientific papers published on this topic (Smith et al,...), there is a risk of about 20% that a response considered complete it is actually not. Non-operated patients should therefore undergo a strict follow-up in the course of which, in case there is a recurrence of disease (recurrence), you run the TME rescue. Even for this approach they have been published many studies that have shown on one hand that wait-and-see approach is safe in patients who achieve a cCR after neoadjuvant therapy; on the other hand, if disease persists, surgery, defined "rescue surgery", leads, in any case, to local control and percentage of OS and DFS completely similar to traditional treatment.

As things stand, there are no studies comparing the two conservative options. The difference between them, based on the results published, are related to the indications: in case of LE, patients are included both with mCR and cCR, whereas wait-and-see approach includes only cCR patients.

This phase II trial is designed to test the hypothesis that conservative treatments, in patients with low-mid rectal cancer who undergo a major or complete clinical response after neoadjuvant treatment, will be safe and effective compared to standard surgery.

Patients will enrol into trial if they will show mCR or cCR at restaging after 7-8 weeks from the end of RT and/or CT; if the response is confirmed at second restaging (11-12 weeks), the patient will be eligible for conservative treatments. If the response is poor after neoadjuvant therapy, seen at first or after second restaging, it is fully recommended to undergo standard surgical treatment.

The investigators will compare rectum-sparing approaches to standard surgery, firstly, in terms of rate of organ preservation at 2 years. Additionally, they will compare survival outcomes (DFS, OS), stoma rates, clinical and tumor factors related to pathological complete response, correlation between major and complete clinical response.

To add value, the investigators will measure quality of life (QoL) in patients treated with rectum-sparing approaches in comparison to patients treated with standard surgery (TME or abdomino-perineal amputation).

The investigators' recent pubblication (Pucciarelli et al, 2013) and experience provide the basis for producing a new multicenter observational trial that can add important information to rectum-sparing approaches in locally advanced rectal cancer patients, highlighting the relationship between neoadjuvant treatment, clinical response and conservative surgical approaches.

Study Design The proposed study is an observational, prospective, multicenter study of patients undergoing neoadjuvant therapy for medium-low rectal cancer.

The investigators opted for an observational study since the Phase 2 study has been completed and Phase 3 studies are objectively, as many Authors report, difficult to perform patients enrollment.

Since this is an observational study that has the aim to evaluate the effectiveness of conservative approaches after neoadjuvant therapy in terms of capacity preservation of organ, they were not given directions on the type of radio and/or chemotherapy treatment. Patients will be enrolled in the study only when patients are candidates (as shown in the studies published on the subject) to a conservative approach. The "registration" of all patients is only meant to evaluate how many patients are potentially candidates for conservative treatment who are undergoing neoadjuvant treatment (secondary endpoint of study). The collection of data concerning the staging of the tumor and basal schemes neoadjuvant therapy aims to identify what type of cancer and what type of neoadjuvant therapy are associated with a higher number of pathological complete responses (secondary endpoint). Finally, for patients who show a cCR, is leaving the ability to run both LE and wait-and-see approach, as the current state, there are no data indicating which option is best in terms of both oncological results and rate of organ preservation.

Study aims

The primary objective of the study is to determine the rate of organ preservation at 2 years in patients with rectal cancer treated with neoadjuvant therapy followed by conservative treatment (LE and wait-and-see). Secondary, the study seeks to:

1. Determine the rate of overall survival (OS), disease-free (DFS) and relapse-free local recurrence at 2, 3, and 5 years after initiation of treatment;
2. Determine the rate of patients without stoma at 2 and at 5 years;
3. Determine the clinical and tumor factors related to treatment and associated with a pathologic complete response (pCR) of the primary tumor;
4. Determine the rate of pCR in patients who are treated with LE and with conventional surgery (TME);
5. Determine the correlation between major or complete clinical response and pCR;
6. Determine the morbidity and mortality after neoadjuvant therapy and conservative approach or TME;
7. Determine the percentage of patients undergoing conservative treatment on total patients running pRT and/or CT;
8. Evaluate the impact of the type of treatment on the ability to perform a preoperative treatment rectum-sparing;
9. Evaluate the impact of surgical approach on bowel function, fecal continence and quality of life (QoL)

Clinical Evaluation and Staging Clinical and pathological primary Tumor, regional Nodes, Metastasis (TNM) stages are determined according to the American Joint Committee on Cancer 7th Edition and for histological grade of adenocarcinoma according to World Health Organization (WHO).

It will be a staging baseline (before any treatment). Patients candidates for pRT and/or CT will be recorded. After the end of pRT and/or CT patients will restage at 7-8 weeks. If there is no evidence of response to therapy, it will proceed to surgery standard (TME), while for patients who show mCR or cCR, there is a second restaging after 11-12 weeks after the end of pRT and/or CT. At the end of this second restaging, the patient will be enrolled in the rectum-sparing protocol if it shows a mCR or cCR, otherwise it will be a candidate for conventional surgery (TME).

Basal clinical staging will be baseline standard for all patients with rectal cancer:

1. digital rectal examination;
2. proctoscopy with rigid endoscope and complete colonoscopy (when it is not executable because the lesion is stenosis, we recommend a double contrast barium enema or colon CT or colonoscopy within 6 months after surgery);
3. pelvic MRI for locoregional staging. If this can not be performed (eg. claustrophobia), it will be accepted pelvic CT or endorectal ultrasound. Lymph nodes with a diameter > 0.5 cm along the short axis will be considered metastatic;
4. chest-abdominal CT for evaluation of distant metastases;
5. carcinoembryonic antigen (CEA) determination;
6. compiling questionnaires (QoL, bowel function, fecal continence).

1st Re-Staging after pRT and/or CT (after 7-8 weeks from the end of radiotherapy):

1. Digital rectal examination;
2. Proctoscopy;
3. chest-abdominal CT;
4. pelvic MRI: if there is evidence of mCR or cCR and the absence of lymph node metastasis on MRI, the patient will be restaged after 11-12 week of the completion of the pRT and/or CT and then treated with rectum sparing approach.

If there is no evidence of mCR or cCR, program surgery (TME) immediately.

2nd Re-staging after pRT and/or CT (after 11-12 weeks from the end of radiotherapy):

1. digital rectal examination;
2. Proctoscopy;
3. pelvic MRI (optional);
4. acquisition of informed consent;
5. Compile questionnaires (QoL, bowel function, fecal continence) optional. If you confirm mCR or cCR, the patient undergoes sparing rectum treatment.

Functional and quality of life assessment As part of the study, they will also be considered bowel function, QoL and fecal continence. Participation in this ancillary study will be voluntary and will cover only those centers that have the ability to manage distribution/collection of the questionnaires.

Functional assessment:

1. MSKCC bowel function instrument.

Quality of life assessment:

1. EORTC QLQ - C30;
2. EORTC QLQ - CR29;
3. Fecal Incontinence Quality of Life scale (FIQL).

Surgical treatment and histopathological exam

Rectal resection with TME This will be carried out according to standard techniques using the open or laparoscopic approach and includes both anterior resection and abdominoperineal rectal resection (Miles procedure).

Local excision This can be done both with traditional technique and with endoscopic technique (TEM, TAMIS, etc.).

The rectum is prepared using standard procedures such as TME approach including prophylactic antibiotics.

For endoscopic techniques it is generally required general anaesthesia, while for LE with a traditional technique is sufficient regional anaesthesia. The patient is positioned in the prone position, lithotomic or side depending on the location of the tumor. Regardless of the technique performed, the following principles should be respected:

1. A gross margin of at least 0.5 cm;
2. full-thickness excision including mucosa, submucosa, muscle and peri-rectal fat;
3. determination of the specimen on the support by pins at the edges in order to facilitate the interpretation of histological pathologist.

The breach on the rectal wall can be closed crosswise with absorbable sutures or it can be left open.

Histological examination

Histological examination must include at least the following information:

1. ypT;
2. Tumor regression grade (TRG) according to the classification of Mandard (see Annex E).

If there is persistence of cancer, at least the following should be described:

1. state of margins;
2. Degree of cellular differentiation;
3. Presence of lymphatic or vascular invasion.

Follow-up Follow-up will be strict, but in any case fall within the patterns of follow-up provided by current national guidelines (see guidelines AIOM follow-up in rectal cancer).

Follow-up after LE or wait- and-see

Patients will be visited every 3 months during the first two years, and then every 6 months in the following three years. For each check, it will be performed:

1. digital rectal examination;
2. Proctoscopy;
3. CEA and routine blood chemistry;
4. MRI every 6 months to 5 years;
5. chest -abdominal CT (annually unless another clinical indication);
6. Colonoscopy (at 1 year, if negative at 3 years, if still negative at 5 years);
7. Compile questionnaires (QoL, bowel function, fecal continence) optional 6 and 12 months after surgery.

Recurrence definition

Recurrences will be distinguished in:

* Local: recurrence in the pelvis, intraluminal or extraluminal;
* Distance: relapse in any other venue. The diagnosis of recurrence will be determined based on clinical, radiological images or biopsy.

Sample size Rectum-sparing approach can be considered clinically acceptable if percentage of conservation of the rectum at two years is not less than 50%.

The collected data on 164 patients who underwent "rectum-sparing" allow to test the hypothesis that the rectum is preserved in 60% of patients with 80% power (exact binomial test for proportions, alpha = 5 %, 1 tail) and the study will be considered positive if it obtains a frequency of conservation of the rectum of not less than 87 cases.

Statistical analysis The analysis results will be reported in accordance with STROBE guidelines (von Elm et al , 2008). For all analyzes, continuous variables are described using the mean and standard deviation of position and appropriate measures when appropriate. Categorical variables will be described using the contingency tables.

Primary endpoint analysis The main analysis will cover the estimated percentage of conservation of the rectum at two years in patients with rectal cancer after pRT and/or CT and "rectum-sparing" treatment.

The percentage of conservation of the rectum will be estimated by the ratio between the number of patients with preservation of the rectum at two years and the total number of patients subjected to local excision or wait- and-see, and reported with 95 % confidence interval.

Analysis of secondary endpoints Secondary analyzes will cover the evaluation of time in the events of death, disease and local recurrence, the description of preoperative treatment, morbidity and frequency of patients without stoma and their association with type of surgery, correlation between mCR or cCR and the pCR, the association between clinical factors and preoperative treatment and surgical and pCR and the impact of the type of surgical treatment on intestinal function, fecal continence and quality of life.

Survival it defines as the time from the date of registration to the event date. In the absence of the event will be considered the date of the last visit. It will be considered events death, local recurrence (recurrence in the pelvis: intraluminal or extraluminal) and distant recurrence (recurrence in any other place). Recurrence diagnosis will be determined based on clinical, radiological images or biopsy.

Survival will be estimated with Kaplan-Meier test. The results will be expressed in terms of survival rates at 2, 3 and 5 years with its 95 % confidence interval. It will also be used a Cox model to estimate the risk of event in the groups of "rectum-sparing" compared to conventional surgery with its 95 % confidence interval.

The frequencies of different treatments administered preoperative, morbidity and packaging of a stoma at 2 and 5 years will be described in terms of percentages and reported with 95 % confidence interval; their association with the type of surgical treatment will be tested by the chi-square test.

The correlation between mCR or cCR and the pCR will be evaluated by estimating the Kappa statistics, which expresses the correlation between the two methods is not due to chance. The results will be expressed with confidence intervals at 95% of bootstrap.

The analysis of factors associated with pCR use a multivariate logistic regression model. It will be used as explanatory variables of clinical information-medical history, the type of preoperative treatment and the type of surgery (TME, LE).

The scales of the questionnaires on intestinal function, fecal continence and quality of life will be built using the standard procedures given in the reference manuals. Mean scores and standard deviations are estimated for each administration of the questionnaires and reported with 95% confidence interval. The trend during the study period will be analyzed using a generalized linear mixed model with a gamma distribution.

ELIGIBILITY:
All patients underwent neoadjuvant therapy for rectal cancer will be registered provided that they satisfy the following requirements:

1. histologically documented adenocarcinoma of the rectum;
2. Up to 12 cm from the anal verge to rectoscopy;
3. Minimum age 18 years old;
4. Able to undergo both neoadjuvant treatment, TME than conservative treatment;
5. For which RT and/or CT fluoropyrimidine ± oxaliplatin or biologic drugs regimens are expected;
6. Able to understand risks and benefits of the protocol.

Criteria for inclusion in the rectum-sparing group (study group):

Of patients registered, they will be eligible for the study rectum-sparing those who have all of the following requirements:

1. Major or complete clinical response at restaging after 7-8 weeks from the end of neoadjuvant therapy, confirmed at second restaging (after 11-12 weeks from the end of neoadjuvant therapy);
2. Written informed consent (after 2nd restaging). Note: They will be subject to wait-and-see approach only patients with cCR.

Criteria of esclusion from protocol:

At restaging after 7-8 weeks and/or after 11-12 weeks, patients who show one of the following characteristics:

1. palpable mass on digital rectal examination;
2. deep ulcer with surface > 2 cm in diameter or obvious signs of endoscopic residual disease;
3. presence of metastatic lymph nodes at MRI (> 5 mm along short axis).

Inclusion criteria to be included to EL or wait- and-see approach:

1. Patients with mCR or cCR at restaging performed after 11-12 weeks after the end of radiotherapy;
2. Ability to understand the protocol;
3. Acquisition of written informed consent.

Inclusion and exclusion criteria to be observed (just follow-up) after LE:

The LE local will be considered as proper treatment if histological assessment will document:

1. ypT0 (cCR);
2. ypT1 but with a TRG degree < 3 and with a differentiation degree of G1-2;
3. histologically margins not involved.

LE will be considered as excessive handling and patients will be advised to undergo TME if histological assessment will document the presence of cancer with at least one of the following characteristics:

1. ypT ≥ 2;
2. Positive margins;
3. TRG ≥ 3;
4. Poor differentiation degree (G3).

Indications to wait-and-see approach This approach, that consists only in observation after neoadjuvant therapy, is reserved only to those patients who show cCR at restaging, as defined previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients underwent neoadjuvant therapy for rectal cancer and have a major or complete clinical response.
  Definitions:
  Major clinical response (mCR) is defined as the absence of:
  • palpable mass at digital rectal exploration, pathological lymph nodes (> 5 mm in diameter along short axis) to pelvic MRI, deep or shallow ulcers > 2 cm in diameter at rectoscopy;
  Clinical complete response (cCR) is defined as the absence of:
  • palpable mass at digital rectal exploration, pathological lymph nodes (> 5 mm in diameter along the short axis) to the pelvic MRI, any endoscopic lesion (a flat scar is considered as absence of endoscopic lesions).
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2016-01; Primary Completion 2021-01 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Rate of organ preservation | 2 years
  The primary objective of th study is to determine the rate of organ preservation at 2 years in patients with rectal cancer treated with neoadjuvant therapy followed by conservative treatment (LE and wait-and-see).

SECONDARY OUTCOMES:
Rate of overall survival (OS) | 2, 3, 5 years
  Rate of overall survival (OS) at 2, 3, and 5 years after initiation of treatment
Rate of disease-free survival (DFS) | 2, 3, 5 years
  Rate of disease-free survival (DFS) at 2, 3, and 5 years after initiation of treatment
Rate of relapse-free local recurrence | 2, 3, 5 years
  Rate of relapse-free local recurrence at 2, 3, and 5 years after initiation of treatment
Rate of patients without stoma | 2, 5 years
  Rate of patients without stoma at 2 and at 5 years
Rate of pCR | At surgery time
  Rate of pCR in patients who are treated with LE and with conventional surgery (TME);
Morbidity | 30 days after surgery
  Morbidity after neoadjuvant therapy and conservative approach or TME
Mortality | 30 days after surgery
  Mortality after neoadjuvant therapy and conservative approach or TME
Rate of patients undergoing conservative treatment | 5 years
  Rate of patients undergoing conservative treatment on total patients running pRT and/or CT
Memorial Sloan-Kettering Cancer Center Bowel Function Instrument | T0: before neoadjuvant treatment; T1: at 10-12 weeks after neoadjuvant treatment; T2: 6 months after T1; T3: 12 months after T1
  MSKCC Bowel Function Instrument (Temple et al., 2005). The questionnaire consists of 18 items that include three subscales (frequency, dietary and urgency/soiling), four individual items of clinical significance ranging (incomplete emptying after a bowel movement, a second bowel movement within 15 min, knowing the difference between gas and bowel movement, inability to control the passage of flatus), and one total score obtained by the sum for all 18 items. Responses to individual items are given on a 5-point Likert scale with the first item (daily frequency of bowel movements) response divided into quintiles. Higher scores indicate better bowel function. The questionnaire has been translated and validated for Italian-speaking patients (Zotti et al., 2011).
Fecal Incontinence Quality of Life Scale | T0: before neoadjuvant treatment; T1: at 10-12 weeks after neoadjuvant treatment; T2: 6 months after T1; T3: 12 months after T1
  FIQL (Rockwood et al., 2000). The questionnaire measures specific quality of life issues expected to affect patients with faecal incontinence. This instrument is composed of 29 items within four domains: lifestyle issues, coping/behaviour, depression/self-perception and embarrassment. The scores range from a minimum score of 1 to a maximum of 4, for all of the scales. The Italian version of the questionnaire has been validated by Altomare et al. (2004).
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 | T0: before neoadjuvant treatment; T1: at 10-12 weeks after neoadjuvant treatment; T2: 6 months after T1; T3: 12 months after T1
  EORTC QLQ-C30 (Aaronson et al., 1993). The questionnaire assesses health status and quality of life of cancer patients using 30 items grouped in one global scale, five multi-item functioning scales (physical, role, social, emotional, and cognitive functions), three symptom scales (fatigue, nausea/vomiting and pain) and six single symptom items (dyspnoea, insomnia, appetite loss, constipation, diarrhoea and financial impact). The items are scored on a four-point Likert scale with higher scores indicating a better level of functioning or a higher level of symptoms. The validity and reliability of the Italian versions of the questionnaire have been established (Apolone et al., 1998).
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Colorectal Cancer Module 29 | T0: before neoadjuvant treatment; T1: at 10-12 weeks after neoadjuvant treatment; T2: 6 months after T1; T3: 12 months after T1
  EORTC QLQ-CR29 (Whistance et al., 2009). The questionnaire measures health-related quality of life in patients with colorectal cancer, using 29 items grouped in four functional scale (body image, anxiety, weight, sex interest men/woman) and 18 symptom scale (urinary frequency, blood and mucus in stool, stool frequency, urinary incontinence, dysuria, abdominal pain, buttock pain, bloating, dry mouth, hair loss, taste, flatulence, fecal incontinence, sore skin, embarrassment, stoma care problems, impotence, dyspareunia). The items are scored on a four-point Likert scale with higher scores indicating a better level of functioning or a higher level of symptoms. The Italian version of the questionnaire is validated and widely used (Whistance et al.,2009).

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Pucciarelli, MD, Principal Investigator — University of Padova
Locations (1):
- Clinica Chirurgica I - Dipartimento di Scienze Chirurgiche, Oncologiche e Gastroenterologiche. Azienda Ospedaliera - Università di Padova, Padua, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barina A, De Paoli A, Delrio P, Guerrieri M, Muratore A, Bianco F, Vespa D, Asteria C, Morpurgo E, Restivo A, Coco C, Pace U, Belluco C, Aschele C, Lonardi S, Valentini V, Mantello G, Maretto I, Del Bianco P, Perin A, Pucciarelli S. Rectal sparing approach after preoperative radio- and/or chemotherapy (RESARCH) in patients with rectal cancer: a multicentre observational study. Tech Coloproctol. 2017 Aug;21(8):633-640. doi: 10.1007/s10151-017-1665-1. Epub 2017 Jul 28. PMID 28755256